CLINICAL TRIAL: NCT00938470
Title: Randomized Phase II Trial of Extended Neoadjuvant Therapy for Locally Advanced Adenocarcinoma of the Esophagus, Gastroesophageal Junction, and Gastric Cardia
Brief Title: Docetaxel, Oxaliplatin, Capecitabine, Fluorouracil, and Radiation Therapy in Treating Patients With Locally Advanced Cancer of the Esophagus or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0849; NCI-2011-01930 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000646724 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Cancer; Gastric Cancer
Keywords: adenocarcinoma of the esophagus; adenocarcinoma of the gastroesophageal junction; stage IIIA gastric cancer; stage IIIB gastric cancer; stage IIIC gastric cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Capecitabine; Docetaxel; Fluorouracil; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (combination chemotherapy, radiation therapy, surgery) (Experimental): Patients receive docetaxel IV over 1 hour and oxaliplatin IV over 2 hours on day 1. Patients also receive capecitabine PO BID on days 1-14. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. After completion of the second course, patients receive fluorouracil IV continuously on days 1-5 and oxaliplatin IV over 2 hours on days 1, 15, and 29. Patients also undergo radiotherapy 5 days a week for 5.5 weeks in the absence of disease progression or unacceptable toxicity. Approximately 4-12 weeks after completion of radiotherapy, patients undergo surgery.
  Interventions: Drug: capecitabine; Drug: docetaxel; Drug: fluorouracil; Drug: oxaliplatin; Radiation: radiation therapy; Procedure: therapeutic conventional surgery
- Arm II (oxaliplatin, fluorouracil, radiation, and surgery) (Active Comparator): Patients receive fluorouracil IV continuously on days 1-5 and oxaliplatin IV over 2 hours on days 1, 15, and 29. Patients also undergo radiotherapy and then surgery as in Arm I.
  Interventions: Drug: fluorouracil; Drug: oxaliplatin; Radiation: radiation therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: capecitabine — Given PO
  Arms: Arm I (combination chemotherapy, radiation therapy, surgery)
Drug: docetaxel — Given IV
  Arms: Arm I (combination chemotherapy, radiation therapy, surgery)
Drug: fluorouracil — Given IV
Drug: oxaliplatin — Given IV
Radiation: radiation therapy — Undergo radiation therapy
Procedure: therapeutic conventional surgery — Undergo surgery

SUMMARY:
This randomized phase II trial studies how well docetaxel, oxaliplatin, capecitabine, fluorouracil, and radiation therapy works compared with fluorouracil when given together with oxaliplatin and radiation therapy in treating patients with cancer of the esophagus or gastroesophageal junction that has spread from where it started to nearby tissue or lymph nodes. Drugs used in chemotherapy, such as docetaxel, oxaliplatin, capecitabine, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving more than one drug (combination chemotherapy) together with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess and compare the pathologic complete response (PCR) rate of patients in Arm A receiving the sequence docetaxel, oxaliplatin, and capecitabine (DOC) followed by 5-fluorouracil (5-FU), oxaliplatin, and radiation therapy (RT) with patients in Arm B receiving only 5-FU, oxaliplatin and RT in patients with potentially resectable adenocarcinoma (ACA) of the esophagus, gastroesophageal junction (GEJ), or gastric cardia.

SECONDARY OBJECTIVES:

I. To assess the adverse event (AE) profile and safety of the proposed treatment in this population.

II. To assess and compare the overall survival (OS) between treatment arms. III. To assess and compare the disease-free survival between treatment arms. IV. To assess and compare the clinical tumor response rate of the proposed regiments when administered before surgery between treatment arms.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive docetaxel intravenously (IV) over 1 hour and oxaliplatin IV over 2 hours on day 1. Patients also receive capecitabine orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. After completion of the second course, patients receive fluorouracil* IV continuously on days 1-5 and oxaliplatin IV over 2 hours on days 1, 15, and 29. Patients also undergo radiotherapy** 5 days a week for 5.5 weeks in the absence of disease progression or unacceptable toxicity. Approximately 4-12 weeks after completion of radiotherapy, patients undergo surgery.

ARM II: Patients receive fluorouracil IV continuously on days 1-5 and oxaliplatin IV over 2 hours on days 1, 15, and 29. Patients also undergo radiotherapy and then surgery as in Arm I.

* NOTE: * Fluorouracil continuous IV infusion begins within 24 hours of radiotherapy and ends within 24 hours of radiotherapy completion.
* NOTE: ** Radiotherapy should begin within 2-6 weeks after completion of 2 courses of docetaxel, oxaliplatin, and capecitabine.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria

* Histological confirmation of adenocarcinoma of the esophagus, gastroesophageal (GE) junction, or gastric cardia
* Tumor must be considered surgically resectable; Note: patients with T4N0M0 tumors that are potentially resectable are also eligible
* Nodal involvement: patients with involvement of celiac nodes, (stations 15-20) are eligible if the primary lesion is mid-thoracic, distal esophagus or GE junction; patients with supraclavicular node involvement are eligible with upper thoracic esophagus primary lesions
* Capable of swallowing pills
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500
* Peripheral platelet count >= 100,000
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper normal limit (UNL)
* Serum glutamic oxaloacetic transaminase (SGOT) (alanine aminotransferase [AST]) =< 3 x UNL
* Creatinine =< 1.5 x UNL
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willingness to return to NCCTG enrolling institution for follow-up
* Patient willing to provide mandatory tissue and blood samples for research purposes
* Patient willing to allow use of FDG PET/CT scans for mandatory research purposes

Exclusion Criteria

* Evidence of distant metastases
* Palpable supraclavicular nodes, biopsy-proven involvement of supraclavicular nodes, or radiographically involved supraclavicular nodes (> 1.5 cm in greatest dimension) for lesions in mid-thoracic, distal thoracic or GE junction
* T1N0M0 or T2N0M0 tumor stage
* Any of the following

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Uncontrolled diabetes (i.e., will interfere with the performance of the FDG PET/CT scans)
* Receiving current treatment or prior treatment for this malignancy
* Other active malignancy 5 years prior to registration, except non-melanotic skin cancer or carcinoma-in-situ of the cervix; if there is a history of prior malignancy, patient must not be receiving other specific treatment (other than hormonal therapy) for cancer
* Prior radiation to > 30% of the marrow cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Alberts, MD, Study Chair — Mayo Clinic
Locations (187):
- United States (187):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Bettendorf, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Luther Midlelfort Hospital, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Yoon HH, Ou FS, Soori GS, Shi Q, Wigle DA, Sticca RP, Miller RC, Leenstra JL, Peller PJ, Ginos B, Heying E, Wu TT, Drevyanko TF, Ko S, Mattar BI, Nikcevich DA, Behrens RJ, Khalil MF, Kim GP, Alberts SR. Induction versus no induction chemotherapy before neoadjuvant chemoradiotherapy and surgery in oesophageal adenocarcinoma: a multicentre randomised phase II trial (NCCTG N0849 [Alliance]). Eur J Cancer. 2021 Jun;150:214-223. doi: 10.1016/j.ejca.2021.03.025. Epub 2021 Apr 29. PMID 33934058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-three participants were enrolled between January 2010 and July 2012.
Pre-assignment Details: Seven participants from arm I were enrolled in the early toxicity evaluation portion. Additional sixty-six participants were randomized to arm I or II on the phase II portion of the study. There were 11 cancellations (5 arm I, 6 arm II) and these participants were excluded in all analyses.
Groups:
- Arm I (DOC, 5FU/O/RT, Surgery): Patients receive 60mg/m^2 docetaxel (D) IV over 1 hour and 85mg/m^2 oxaliplatin (O) IV over 2 hours on day 1. Patients also receive 625 mg/m^2/dose twice a day of capecitabine (C) PO BID on days 1-14. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. After completion of the second course, patients receive 180 mg/m^2 per day of fluorouracil (5FU) IV continuously on days 1-5 and 85 mg/m^2 oxaliplatin (O) IV over 2 hours on days 1, 15, and 29. Patients also undergo radiation therapy (RT) 5 days a week for 5.5 weeks in the absence of disease progression or unacceptable toxicity. Approximately 4-12 weeks after completion of radiation therapy, patients undergo surgery.
- Arm II (5FU/O/RT, Surgery): Patients receive 180 mg/m^2 per day of fluorouracil (5FU) IV continuously on days 1-5 and 85 mg/m^2 of oxaliplatin (O) IV over 2 hours on days 1, 15, and 29. Patients also undergo radiation therapy (RT) and then surgery.
Period: Overall Study
Arm/Group | Arm I (DOC, 5FU/O/RT, Surgery) | Arm II (5FU/O/RT, Surgery)
Started | 34 | 28
Completed | 27 | 25
Not Completed | 7 | 3
Not completed — Disease Progression | 3 | 0
Not completed — Alternate Treatment | 1 | 0
Not completed — Death | 3 | 2
Not completed — Other Reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible randomized participants who initiated first cycle of protocol treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (DOC, 5FU/O/RT, Surgery) | Arm II (5FU/O/RT, Surgery) | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Median (Full Range); unit: years] | 62.5 [38 to 78] | 65 [44 to 88] | 63 [38 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 23 | 23 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 27 | 55
ECOG Performance Status 0-1 [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status:
  0=Asymptomatic and fully active
  1=Symptomatic and fully ambulatory
  Participants | 28 | 27 | 55
Tumor Stage [Count of Participants; unit: Participants] — Staging group was defined by primary tumor (T), regional (N) and distant metastasis (M).
  II= T2N0M0, T3N0M0 or T1-2, N1M0; III= T1-2,N2M0 or T3N1M0, T4aN0M0 or T3N2M0 or T4a,N1-2, M0 or T4b, Any N, M0 or Any T, N3, M0
  M0=No M N0=No N M N1=M in 1-2 N N2=M in 3-6 N N3=M in >=7 N NX=N cannot be assessed (NA) T1=Invades lamina propria, muscularis mucosae, or submucosa T2=Invades muscularis propria T3=Invades adventitia T4=Invades adjacent structures T4a=Resectable T invading pleura, pericardium, or diaphragm T4b=Unresectable T invading other adjacent structures TX=T NA
  Participants
    II | 6 | 9 | 15
    III | 22 | 18 | 40
Site of Tumor [Count of Participants; unit: Participants]
  Esophagus | 16 | 11 | 27
  Gastroesophageal Junction | 12 | 14 | 26
  Gastric Cardia | 0 | 2 | 2
Measurable Disease [Count of Participants; unit: Participants]
  Yes | 11 | 11 | 22
  No | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathologic Complete Response (PCR)
Description: Pathologic complete response was defined as no gross or microscopic tumor identified with the surgical specimen. All lymph nodes should be free of tumor to document a PCR. If no gross tumor is visible, section around the area of inflammation (nodularity) should be made every 2-3 cm and specimens examined.
Time Frame: Up to 2 years
Population: Eligible randomized participants who initiated first cycle of protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (DOC, 5FU/O/RT, Surgery) | Arm II (5FU/O/RT, Surgery)
Number analyzed (Participants) | 28 | 27
percentage of participants | 28.6 [13.2 to 48.7] | 40.7 [22.4 to 61.2]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to the time of death from any cause. Overall survival was censored at the date of last follow-up visit for patients who are still alive or loss of follow-up.
Time Frame: Up to 2 years
Population: Eligible randomized participants who initiated first cycle of protocol treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (DOC, 5FU/O/RT, Surgery) | Arm II (5FU/O/RT, Surgery)
Number analyzed (Participants) | 28 | 27
months | NA [24.0 to NA] — Median survival and upper limit of 95% CI are not attainable. | 18.8 [13.3 to NA] — Upper limit of 95% CI is not attainable.

3. Secondary Outcome: Disease-free Survival
Description: Disease-free survival was defined as the time from randomization to the date of recurrent or death, whichever comes first.
Time Frame: Up to 2 years
Population: Eligible randomized participants who initiated first cycle of protocol treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (DOC, 5FU/O/RT, Surgery) | Arm II (5FU/O/RT, Surgery)
Number analyzed (Participants) | 28 | 27
months | 31.2 [15.4 to NA] — Upper limit of 95% CI is not attainable. | 17.0 [11.1 to NA] — Upper limit of 95% CI is not attainable.

4. Secondary Outcome: Number of Participants Who Experienced a Maximum Grade of 3 or Above Adverse Event
Description: Adverse events were assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 2 years
Population: Eligible randomized participants who initiated first cycle of protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (DOC, 5FU/O/RT, Surgery) | Arm II (5FU/O/RT, Surgery)
Number analyzed (Participants) | 28 | 27
Participants
  Grade 3=Severe | 10 | 12
  Grade 4=Life threatening | 10 | 7
  Grade 5=Death | 4 | 4

5. Secondary Outcome: Percentage of Participants With Overall Clinical Tumor Response (CR or PR)
Description: Overall clinical tumor response rate was defined as the percentage of evaluable participants who achieved either complete response (CR) or partial response (PR) noted on the objective status from pre-surgical staging (for arm II) or either from pre-RT or pre-surgical staging (for arm I).> CR was defined as disappearance of all non-target lesion (TL) and normalization of tumor biomarker level, all lymph nodes (LN) must be non-pathological in size (<1 cm short axis); or disappearance of all TL and normalization of tumor biomarkers, any pathological LN (whether target or non-target) must have reduction in short axis to <1 cm; or >=30% decrease in the sum of the diameters of TL taking as reference the baseline sum of the diameters.
Time Frame: Up to 2 years
Population: Eligible randomized participants who initiated first cycle of protocol treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (DOC, 5FU/O/RT, Surgery) | Arm II (5FU/O/RT, Surgery)
Number analyzed (Participants) | 28 | 27
percentage of participants | 32.1 [15.9 to 52.4] | 33.3 [16.5 to 54.0]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events data were reported on 55 eligible randomized participants who initiated first cycle of protocol treatment, 1 ineligible Arm II participant and 6 eligible Arm I participants who enrolled onto the early toxicity evaluation portion of the study.
Arm/Group | Arm I (DOC, 5FU/O/RT, Surgery) | Arm II (5FU/O/RT, Surgery)
Serious Adverse Events (participants affected / at risk) | 7/34 | 7/28
Other Adverse Events (participants affected / at risk) | 34/34 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (DOC, 5FU/O/RT, Surgery) (N=34) | Arm II (5FU/O/RT, Surgery) (N=28)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Death NOS (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (DOC, 5FU/O/RT, Surgery) (N=34) | Arm II (5FU/O/RT, Surgery) (N=28)
Anemia (Blood and lymphatic system disorders) | 7 (10) | 8 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (3)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 21 (41) | 15 (22)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 26 (68) | 22 (41)
Esophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Esophagitis (Gastrointestinal disorders) | 3 (3) | 6 (6)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (3) | 2 (2)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 30 (83) | 24 (44)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 21 (35) | 18 (32)
Edema limbs (General disorders) | 2 (2) | 1 (1)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 15 (28) | 11 (14)
Fever (General disorders) | 2 (2) | 2 (2)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Bone infection (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (5) | 2 (2)
Lung infection (Infections and infestations) | 2 (3) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Gastric anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (5) | 0 (0)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 4 (5) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 3 (4)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (5) | 9 (14)
Neutrophil count decreased (Investigations) | 28 (47) | 5 (5)
Platelet count decreased (Investigations) | 22 (66) | 22 (43)
Weight loss (Investigations) | 8 (20) | 8 (12)
White blood cell decreased (Investigations) | 28 (74) | 13 (20)
Anorexia (Metabolism and nutrition disorders) | 8 (10) | 11 (12)
Dehydration (Metabolism and nutrition disorders) | 7 (9) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6) | 5 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (8) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (4) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (59) | 18 (24)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (5) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (44) | 13 (19)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (13) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 3 (9) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less